CLINICAL TRIAL: NCT00918424
Title: Long Term Multiple Dose, Open-Label, Multi-Center Study to Evaluate the Safety and Tolerability of OXC XR as Adjunctive Therapy in Pediatric Subjects With Refractory Partial Epilepsy
Brief Title: Long Term Study of the Safety of OXC XR as in Pediatric Epilepsy Subjects
Status: Approved for marketing | Type: Expanded Access
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 804P303
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine Extended Release — OXC XR is a once-daily formulation of oxcarbazepine and is given at the same dosage levels.
  Other Names: Oxtellar XR

SUMMARY:
Follow-on study to continue evaluation of the safety of OXC XR as adjunctive therapy in pediatric epilepsy

DETAILED DESCRIPTION:
Pediatric patients with partial onset epilepsy enrolled in a pharmacokinetic study of OXC XR were allowed to continue treatment with the investigational drug in this extensión study. The primary interest was in assessing the safety of treatment with OXC XR over a period of months.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed assent (IAF), as appropriate, with written informed permission (and informed consent (ICF) where required by regional laws or regulations) from the parent or legally-authorized representative (LAR).
2. Was eligible for and completed the 804P107 study.
3. Weight within the 25 - 75 % weight-for-age percentiles based on the National Center for Health Statistics Growth Charts, and not less than 15.0kg, when entering the 804P107 study.
4. Able and willing to swallow whole tablets.
5. Females of childbearing potential (FOCP) should either be sexually inactive (abstinent) for 14 days prior to entering the 804P107 804P107, throughout this study, and for four days following the last dose; or, if sexually active, will be using one of the following acceptable birth control methods:

   1. Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) six months minimum;
   2. Intrauterine device in place for at least three months;
   3. Barrier methods (condom, diaphragm) with spermicide for at least 14 days prior to the first dose of the 804P107 study, throughout the study, and for four days following the last dose;
   4. Surgical sterilization of the partner (vasectomy for six months minimum);
   5. Hormonal contraceptives in addition to a barrier method (condom, diaphragm) with spermicide for at least 14 days prior to the first dose of the 804P107 study, throughout the study, and for four days following the last dose.

Exclusion Criteria:

1. Meets criteria for history of major depressive or manic episode, according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Text Revision.
2. Any history of suicide intent and/or attempt.
3. History or presence of clinically significant, chronic medical condition, especially those contraindicating antiseizure medication, (e.g., any neurological, gastrointestinal, endocrine, cardiovascular, pulmonary, hematological, immunologic, renal, hepatic or metabolic disease) that may affect the safety of the subject in the opinion of the Investigator.
4. Use of felbamate with less than 18 months of continuous exposure prior to screening for the 804P107 study and continuous use throughout this study.
5. Frequent need of rescue benzodiazepines (more than once in a 28 day period).
6. Use of diuretics or other sodium-lowering medications.
7. History or presence of clinically significant laboratory, electrocardiogram (ECG), or vital sign abnormalities that may affect the safety of the subject, in the opinion of the Investigator at the end of study visit for the 804P107 study.
8. Presence of potential hepatic function impairment as shown by, but not limited to, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal (ULN), or total bilirubin >1.5 times ULN, according to the lab results of the 804P107 study.
9. Presence of suspected impairment of renal function defined by serum creatinine ≥1.5 times ULN, according to the lab results of the 804P107 study.
10. Females who are pregnant or lactating.
11. Previous known hypersensitivity to OXC or other related drugs, such as carbamazepine.
12. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2009-06

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Site 03, Loxahatchee Groves, Florida
  - Palm Beach, Florida
  - Site 02, Rockville, Maryland
  - Site 05, Rochester, New York
  - Kingsport, Tennessee
  - Site 07, San Antonio, Texas